CLINICAL TRIAL: NCT06193122
Title: Investigation of Three-Dimensional Ultrasound and Spectroscopy as Early Indicators of Breast Cancer Response to Neoadjuvant Treatment
Brief Title: Three-Dimensional Ultrasound and Spectroscopy as Early Indicators of Breast Cancer Response to Neoadjuvant Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Radiation Oncologist and Clinical Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 5552
Record Dates: First submitted 2023-12-08; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant Chemotherapy; Three-Dimensional Ultrasound; Spectroscopy
MeSH Terms: conditions — Breast Neoplasms | interventions — Spectrum Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard neoadjuvant treatments: Patients will be assessed using ultrasound imaging 3D and spectroscopy at the following intervals: once immediately prior to commencing neoadjuvant treatment. Once treatment begins, patients will be imaged at weeks 2, 4, 8, 12 and then prior to their surgery.
  Interventions: Device: Ultrasound imaging 3D and Spectroscopy

INTERVENTIONS:
Device: Ultrasound imaging 3D and Spectroscopy — Ultrasound imaging and spectroscopy will consist of collecting three dimensional data. Regions of interest in each of the tumour images and in the adjacent normal tissue will be selected for analysis.

SUMMARY:
The purpose of the study is to test the hypothesis that ultrasound imaging and spectroscopy may be used as a predictive marker of advanced tumour response to neoadjuvant treatment consisting of chemotherapy or concurrent chemotherapy-radiotherapy. The main goal is to select the best ultrasound spectroscopy parameter and vascular-distribution index to use as an early predictor of pathological complete or partial response as a primary endpoint and tumour size decrease as a secondary endpoint.

DETAILED DESCRIPTION:
This project is an early validation study in human subjects that will use three-dimensional ultrasound imaging and spectroscopy to monitor cell death occurring at various time points during a patient's treatment for advanced breast cancer. Standard neoadjuvant treatments for breast cancer consisting of combined chemotherapy and radiotherapy will be used in patients. Reponses will be followed with ultrasound imaging and spectroscopy at regular predetermined time-points. The research is exploratory since upon data analysis it will examine the use of different ultrasound backscatter parameters as potential markers of cell death and correlate these with changes in tumour size and complete pathological response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed breast carcinoma, stage I-IV, which has not been treated with any first-line therapy and will be treated with neoadjuvant chemotherapy or neoadjuvant combined chemo-radiotherapy.
2. Disease must be measurable by ultrasound, or MRI performed within 28 days prior to treatment.
3. Eastern Co-operative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Life expectancy of at least 6 months.
5. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to dosing:

   (i) hemoglobin >90 mg/dL (ii) leukocytes >3,000/mL (iii) absolute neutrophil count >1,500/mL (iv) platelets >100,000/mL (v) total bilirubin within normal institutional limits (vi) AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal (vii) creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional upper limit of normal.
6. Patients should have the ability to understand and the willingness to sign a written informed consent document. Signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

1. Chemotherapy, radiotherapy, or major surgery within 4 weeks prior to registering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to registration.
2. Receiving any other investigational agents.
3. Known brain metastases.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition.
5. Contraindications to radiotherapy such as but not limited to:

   (i) previous radiotherapy to an involved area (ii) active collagen vascular disease (iii) genetic diseases associated with hyper-radiosensitivity.
6. Any clinically serious infections requiring systemic anti-bacterial, antifungal or antiviral therapy.
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, and cardiac arrhythmia.
8. Psychiatric illness/social situations that would limit compliance with study requirements.
9. History of active ongoing seizure disorder.
10. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
11. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and women and members of all races and ethnic groups who will receive standard Neoadjuvant treatment for Breast Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Ultrasound imaging and spectroscopy as a predictive marker of early predictor of complete pathological response. | Up to 5 years
  The primary endpoint of this study will be to correlate changes in ultrasound backscatter parameters obtained throughout the course of treatment with complete or partial pathological response.

SECONDARY OUTCOMES:
To Examine the change in tumour size over the course of treatment and correlating it to changes in ultrasound backscatter parameters. | Up to 5 years
  Tumour size will be measured using conventional B-mode ultrasound imaging. Both the tumour's maximum dimensions length, width, and height in cm will be considered.
To Examine the change in tumour Volumen over the course of treatment and correlating it to changes in ultrasound backscatter parameters. | Up to 5 years
  The Volumen of the tumor will be measured by conventional ultrasound in B mode. The volume of the tumor in cm3 will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Czarnota, PhD, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No